CLINICAL TRIAL: NCT04650594
Title: Clinical Results, Isokinetic Analysis and Radiologic Outcomes of Knee MUTARS Protheses Replacement for Malignant Tumours of Bone
Brief Title: Functional Outcomes of Knee Protheses for Malignant Tumours of Bone
Acronym: ISOMUTAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator's decision
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019_60; 2020-A01796-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-05

CONDITIONS: Knee Disease; Bone Cancer
Keywords: Tumour; prosthese replacement; functional outcomes; knee; isokinetic
MeSH Terms: conditions — Bone Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- case group (Experimental): Patients with knee bone malignancy
  Interventions: Procedure: MUTARS® modular reconstruction prostheses

INTERVENTIONS:
Procedure: MUTARS® modular reconstruction prostheses — Patients with MUTARS® modular reconstruction prostheses following primary or secondary knee bone malignancy with minimal follow-up of one year

SUMMARY:
The placement of mega knee prosthesis is a necessity after a large tumor resection and oncological. These mega knee prostheses implanted in the context of oncological surgery have been very few evaluated in the literature.

Active knee extension is essential in order to walk properly. The study propose the evaluation of this prosthesis by checking the possibility of locking of the prosthetic joint and thus the possibility of active walking.

A more in-depth, isokinetic analysis at 1 year of follow-up will also be done in an exploratory manner, as the literature has no data on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Patient with MUTARS® modular reconstruction prostheses following primary or secondary knee bone malignancy with minimal follow-up of one year,
* Cardiological follow-up including at least one ECG and a clinical examination of less than 1 year (ability to perform the isokinetic test),
* Written informed consent from patient,
* Socially insured patient,
* Patient willing to comply with all study procedures and study duration.

Exclusion Criteria:

* - Underage,
* Less than a one-year follow-up after surgery (stability of results is not achieved if follow-up is less than one year),
* Meniscal lesion knee healthy side,
* Prosthetic surgery of the knee healthy side,
* Patient with an unbound fracture,
* Patient without cardiological follow-up,
* Pregnant or breastfeeding woman,
* Inability to receive information, consent and participate in the whole study,
* No social insurance cover,
* No written consent,
* Person under judicial protection or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
Rate of patients with active locking of the operated knee | Baseline
  rate of patients with successful locking will be estimated by the frequency observed Active locking of the operated knee

SECONDARY OUTCOMES:
Measurement of joint amplitudes | Baseline
  Functional results of patients with medullary reconstruction prosthesis,joint amplitudes in flexion-extension and in active, passive,
Presence of frontal and sagittal laxity | Baseline
  Functional results of patients with medullary reconstruction prosthesis
Musculoskeletal Tumour Society Scoring System (MSTS) | Baseline
  The MSTS Score may be used as a functional measure for patients with sarcoma involving the upper limb. The score includes 6 measures (pain, function, emotional acceptance, hand position, manual dexterity, lifting ability) each measure with a maximum of 5 points. The maximum overall score is 30 points. The score is designed to be used after the procedure and is therefore only collected post-operatively.
Oxford knee score | Baseline
  The Oxford Knee Score (OKS) is a Patient Reported Outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty.
  Each of the 12 answers are assigned the previously defined number of points. They range from 1 = least difficult to 5 = most difficult. The 12 ratings are then added together to give a total score used to assess the patient.
  Functional results of patients with medullary reconstruction prosthesis
KOOS for the daily impact (subjective score) | Baseline
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient-reported outcome measurement instrument, developed to assess the patient's opinion about their knee and associated problems Functional results of patients with medullary reconstruction prosthesis
International Knee Society (IKS) score | Baseline
  International Knee Society score : range 0 to 200, a higher score means a better outcome Functional results of patients with medullary reconstruction prosthesis
Radiological evaluation | Baseline
  Radiological results of patients with medullary reconstruction prosthesis Radiological criterion : Lower limb axis,Blackburn and Peel index for patellar height, Radiological signs of loosening
Isokinetic strength of the quadriceps and ischio-leg muscles during knee flexion and extension by isokinetic machine type Contrex®. | Baseline
  Muscle recovery of the operated limb compared to the healthy limb
The test angular velocities are 60°/s and 180°/s in concentric contraction mode by isokinetic machine type Contrex®. | Baseline
  Muscle recovery of the operated limb compared to the healthy limb
  .

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Szymanski, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Swynghedauw, Lille, France